CLINICAL TRIAL: NCT07322952
Title: Randomized Controlled Trial of a Gamified Tai Chi Intervention to Improve Executive Function in Children With Autism Spectrum Disorder
Brief Title: Gamified Tai Chi Intervention to Improve Executive Function in Children With Autism Spectrum Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan University Guangzhou (Other)
Collaborators: Chaozhou Special Education School (Unknown)
Responsible Party: Principal Investigator, Ma Ruisi, Lecturer, School of Physical Education, Jinan University, Jinan University Guangzhou
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025LCLL-141
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder (ASD
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants will maintain their routine rehabilitation courses and standard physical education classes as per the school curriculum. No additional Tai Chi training will be provided during the 12 months study period. They may be offered Tai Chi training after the study conclusion (Waitlist design).
- Traditional Tai Chi Group (Active Comparator): Participants will receive a 12 months standard Traditional Tai Chi training (3 sessions/week, 45 mins/session). This group performs the same physical movements as the experimental group but without any gamification, scoring systems, or interactive game scenarios.
  Interventions: Behavioral: Traditional Tai Chi Group
- Gamified Tai Chi Group (Experimental): Participants will receive a 12 months Gamified Tai Chi intervention (3 sessions/week, 45 mins/session). The intervention integrates the MDA (Mechanics, Dynamics, Aesthetics) framework and exergaming elements into traditional Tai Chi movements to target executive functions.
  Interventions: Behavioral: Gamified Tai Chi Program

INTERVENTIONS:
Behavioral: Gamified Tai Chi Program — Participants will receive a 12 months Gamified Tai Chi intervention (3 sessions/week, 45 mins/session). The intervention integrates the MDA (Mechanics, Dynamics, Aesthetics) framework and exergaming elements into traditional Tai Chi movements to target executive functions.
  Arms: Gamified Tai Chi Group
Behavioral: Traditional Tai Chi Group — Participants will receive a 12 months standard Traditional Tai Chi training (3 sessions/week, 45 mins/session). This group performs the same physical movements as the experimental group but without any gamification, scoring systems, or interactive game scenarios.
  Arms: Traditional Tai Chi Group

SUMMARY:
This randomized controlled trial evaluates the effectiveness of a "Gamified Tai Chi" intervention on improving executive functions (such as inhibitory control, working memory, and cognitive flexibility) in children with Autism Spectrum Disorder (ASD).

The study aims to determine whether integrating game mechanics (based on the Mechanics, Dynamics, and Aesthetics framework) into Tai Chi training offers superior benefits compared to traditional Tai Chi training or routine care.

Approximately 200 children aged 8-15 years will be randomly assigned to one of three groups for a 12 months period:

Gamified Tai Chi Group: Participants will attend sessions combining simplified Tai Chi forms with interactive tasks, such as digital chasing games and cooperative challenges, using a point-based reward system to enhance engagement.

Traditional Tai Chi Group: Participants will learn the same Tai Chi movements but via standard instruction methods without gamification elements.

Control Group: Participants will continue their routine rehabilitation or physical education classes (Waitlist design).

Assessors who are blinded to group allocation will evaluate outcomes at baseline and post-intervention using standardized cognitive tasks (e.g., Flanker task, 1-back task) and behavioral questionnaires regarding social functioning and daily living skills.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 15 years at enrollment.
* Clinical diagnosis of autism spectrum disorder based on DSM Fifth Edition or ICD Eleventh Revision, confirmed by a qualified child psychiatrist or psychologist.
* Basic receptive and expressive language abilities sufficient to understand simple verbal instructions and to express basic needs.
* Ability to participate in group based physical activities as judged by clinicians or teachers.
* Written informed consent provided by a legal guardian and assent provided by the child within his or her level of understanding.

Exclusion Criteria:

* Coexisting severe psychiatric disorders such as psychotic disorders or major mood disorders, or intellectual disability with an intelligence quotient less than 70.
* Uncontrolled epilepsy, or medical conditions that may compromise exercise safety, including but not limited to significant cardiovascular disease, respiratory disease, or musculoskeletal disorders.
* Receipt of systematic interventions specifically targeting executive function or regular martial arts or Tai Chi training during the three months prior to enrollment.
* Inability to follow verbal instructions, or marked behavior problems that make participation in group activities unsafe or infeasible, as judged by clinicians or teachers.
* Any other condition that the research team considers likely to interfere with participation in the intervention or with outcome assessment.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 223 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in working memory measured by 1 back task accuracy | Change from baseline to 6 months after randomization
  Working memory will be assessed with a computerized 1 back task. The primary outcome will be mean accuracy across all experimental trials. Higher scores indicate better working memory performance.
Change in inhibitory control measured by Flanker task accuracy | Change from baseline to 6 month after randomization
  Inhibitory control will be assessed with a child friendly computerized Flanker task. The primary outcome will be mean accuracy on incongruent trials. Higher scores indicate better inhibitory control.
Change in cognitive flexibility measured by More Odd Shifting task accuracy | Change from baseline to 6 months after randomization
  Cognitive flexibility will be assessed with a computerized More Odd Shifting task that requires switching between judging number magnitude and number parity. The primary outcome will be mean accuracy on mixed blocks that require task switching. Higher scores indicate better cognitive flexibility.

SECONDARY OUTCOMES:
Change in social responsiveness measured by the Social Responsiveness Scale-Second Edition (SRS-2) | Change from baseline to 6 months after randomization
  Social functioning will be assessed using the caregiver rated Social Responsiveness Scale-Second Edition (SRS-2). The primary outcome for this measure will be the SRS-2 total T score. Higher scores indicate more severe social communication and interaction difficulties.
Change in functional independence in daily living measured by the WeeFIM | Change from baseline to 6 months after randomization
  Activities of daily living will be evaluated with the Functional Independence Measure for Children (WeeFIM). The outcome will be the WeeFIM total score summarizing self care, mobility and cognition items. Higher scores indicate greater functional independence in everyday life.
Change in behavior problems measured by the Child Behavior Checklist for ages 6-18 (CBCL/6-18) | Change from baseline to 6 months after randomization
  Behavior problems will be assessed using the parent rated Child Behavior Checklist for ages 6-18 (CBCL/6-18). The main outcomes will be T scores on attention related and hyperactivity related scales. Higher T scores indicate more severe behavior problems.
Change in autism symptom severity measured by the Childhood Autism Rating Scale (CARS) | Change from baseline to 6 months after randomization
  Autism symptom severity will be assessed using the Childhood Autism Rating Scale (CARS). The outcome will be the CARS total score based on clinician ratings across core symptom domains. Higher scores indicate more severe autism related symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaozhou Special Education School, Chaozhou, Gaungdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this trial involves a small sample of children with autism spectrum disorder, who are considered a vulnerable population. Given the risk of re identification in this specific clinical and educational setting, and according to the requirements of the ethics committee and the consent obtained from legal guardians, only de identified aggregate results will be reported and shared.